CLINICAL TRIAL: NCT03825822
Title: A Cluster Randomized Clinical Trial to Evaluate the Effectiveness of a Multifaceted Knowledge Translation Intervention in Hospitalized Infants: the Implementation of Infant Pain Practice Change (ImPaC) Resource
Brief Title: The Effectiveness of a Multifaceted Knowledge Translation Intervention on Pain in Hospitalized Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Bonnie Stevens, Senior Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REB1000061599
Record Dates: First submitted 2019-01-25; First posted 2019-01-31 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Pain; Infant
Keywords: Pain; Procedures; Infants; Assessment; Management; Knowledge translation; Context; Implementation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding will only be possible for the data analysts because no identifiable information about the sites, including the infants in the NICUs, will be available in the database or data extracted from the database. The code associating units with the data will be securely stored by the lead site, kept separate from the data, and only made available to the lead site Research Team for analyses purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ImPaC Resource Intervention (INT) (Experimental): The INT arm will receive the 7-step web-based ImPaC intervention to use over 6 months. The intervention is divided into the Plan Stage and the Change Stage. The Plan Stage (steps 1-4) is expected to be completed in 1 month. The Change Stage (steps 5-7) is expected to be completed in 1-2 months. We anticipate that Change Teams will be able to complete 2 cycles of change over the 6-month intervention period.
  Interventions: Behavioral: ImPaC Resource Intervention (INT)
- Standard Practice (SP) (Other): The SP arm will continue as usual with their unit or institutional standard pain practices and any strategies that they would normally use to improve them (e.g. new staff orientation).
  Interventions: Other: Standard Practice (SP)

INTERVENTIONS:
Behavioral: ImPaC Resource Intervention (INT) — A Change Team will lead the implementation process of the ImPaC Resource using the steps:
  Step 1: Complete a checklist to ensure its members can commit to responsibilities.
  Step 2: Reflect on the unit's readiness for change.
  Step 3: Perform an audit on 10 to 15 medical charts.
  Step 4: Identify a practice change based on audit results (pain assessment or pain treatment). Develop an aim statement for the practice change.
  Step 5: Select the KT strategies and plan the implementation.
  Step 6: Perform an audit on 10 to 15 medical charts.
  Step 7: Examine the effectiveness of the implementation and decide on the aim and KT strategies for the next cycle of change.
  Arms: ImPaC Resource Intervention (INT)
Other: Standard Practice (SP) — The SP arm will continue as usual with their standard pain practices and will be offered the intervention 6 months after randomization and completion of data collection.
  Arms: Standard Practice (SP)

SUMMARY:
Hospitalized infants undergo multiple painful procedures daily. Despite generation of a significant amount of evidence, procedural pain assessment and management in infants continues to be suboptimal. Untreated pain at this vital developmental juncture is associated with negative behavioural and neurodevelopmental consequences. To address this knowledge to practice gap, the investigators developed the Implementation of Infant Pain Practice Change (ImPaC) Resource (Resource) to guide change in health care professionals' pain practice behaviour.

The aim of this study is (i) to evaluate the clinical effectiveness of the Resource (primary), (ii) to evaluate the implementation effectiveness of the Resource (secondary), and (iii) to explore how organizational context influences clinical and implementation outcomes (other).

Eighteen Level 2 or Level 3 Neonatal Intensive Care Units (NICUs) with a minimum of 15 beds across Canada will be included in a cluster randomized controlled trial (RCT). The NICUs will be randomized following baseline data collection using a computer-generated random allocation sequence (randomize.net) to either the intervention (INT) or standard practice (SP) arms. Those in INT arm will receive the Resource for a 6-month period. NICUs in the SP arm will continue as usual with their unit or institutional pain practices. They will be offered the Resource following outcomes assessment. Clinical outcomes will be assessed six months after randomization. Primary clinical outcomes include (1) the proportion of infants in the NICU who have procedural pain assessed with a valid pain measure, (2) the proportion of infants in the NICU who have procedural pain managed with an evidence-based pharmacological or physical intervention, and (3) the total number of painful procedures per infant in the NICU. Implementation outcomes will include feasibility, fidelity, cost, and reach. Organizational context will be assessed by using the Alberta Context Tool.

ELIGIBILITY:
NICUs in pediatric or general hospitals will be invited to participate in this study if they:

* are Level 2 or Level 3 NICUs in Canada,
* have at least 15 beds, and
* agree to participate for 24 months.

Infants' clinical charts data will be collected if infants:

• are hospitalized for the designated 24h period for chart review,

Infants' charts will be excluded if:

* infant leaves the unit at any time (transfer, surgeries, procedures) during the designated 24h period for chart review,
* parents request to opt out of the study.

Staff members of the NICU will be eligible to participate on the ImPaC change team if they:

* are a health care professional,
* are English speaking,
* have 3+ years of experience in the NICU,
* have flexibility within their role to engage in the study, and
* have leadership experience (e.g. in an advanced practice or clinical role). There is no exclusion criteria.

Staff members of the NICU will be invited to complete the organizational context survey if they:

* have 6 months experience in the NICU, and
* work 0.5 FTE or above. There is no exclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Proportion of infants with procedural pain assessed | At 6 months after randomization
  The proportion of infants in the NICU who have procedural pain assessed with a valid pain measure documented on clinical charts over a standardized 24-hour period.
Proportion of infants with procedural pain management | At 6 months after randomization
  The proportion of infants in the NICU who have procedural pain managed with evidence-based pharmacological or physical interventions documented on clinical charts over a standardized 24-hour period.
Frequency of painful procedures | At 6 months after randomization
  Total number of painful procedures (e.g. heel lance, arterial puncture, eye examination) per infant in the NICU documented in clinical charts over a standardized 24-hour period.

SECONDARY OUTCOMES:
Use of the Resource (Feasibility/Fidelity) | At completion of 6-month intervention for INT arm
  Feasibility and fidelity will be measured using Resource metrics that address (a) if all 7 steps of the Resource are completed (feasibility) and (b) if all the 7 steps are completed as intended in order (fidelity). Feasibility and fidelity metrics (data captured from the backend of the Resource website) will be electronically collected at the end of the 6-month implementation of the intervention. There is no specific measure to assess feasibility or fidelity.
Implementation costs | At completion of 6-month intervention for INT arm
  Implementation costs will be assessed in terms of (a) incidental costs (Canadian dollars) associated with knowledge translation and implementation activity (e.g., printing posters, refreshments for education sessions) documented in the Resource; and (b) time (hours/minutes) spent by each member of the Change Team in completing each step of the Resource. Time will be converted to actual costs by multiplying hours spent by the hourly wage of the Change Team members. Data will be captured from Resource metrics (data captured from the backend of the website) at the end of the 6-month implementation of the intervention. There is no specific measure to assess reach.
Integration of the Resource into the practice (Reach) | At completion of 6-month intervention for INT arm
  Number of providers in the NICU who receive each knowledge translation and implementation activity that will be documented in the Resource website by the Change Team members. Data will be captured from the Resource website at the end of the 6-month implementation of the intervention. There is no specific measure to assess reach.

OTHER OUTCOMES:
Context evaluation (ACT) | Baseline
  Local context characteristics will be assessed with the Alberta Context Tool completed by staff nurses.
Context evaluation (ACT) | Prior to start of intervention for INT arm
  Local context characteristics will be assessed with the Alberta Context Tool completed by Change Team members.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Stevens, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooke, J. (2013). SUS: A Retrospective. Journal of Usability Studies, 8(2), 29-40. https://doi.org/10.1074/jbc.R115.675280
- [Background] Brooke, J. (1996). SUS - A quick and dirty usability scale. Usability Evaluation in Industry, 189(194), 4-7. https://doi.org/10.1002/hbm.20701
- [Background] Cruz MD, Fernandes AM, Oliveira CR. Epidemiology of painful procedures performed in neonates: A systematic review of observational studies. Eur J Pain. 2016 Apr;20(4):489-98. doi: 10.1002/ejp.757. Epub 2015 Jul 29. PMID 26223408
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Estabrooks CA, Squires JE, Cummings GG, Birdsell JM, Norton PG. Development and assessment of the Alberta Context Tool. BMC Health Serv Res. 2009 Dec 15;9:234. doi: 10.1186/1472-6963-9-234. PMID 20003531
- [Background] Forman, J., & Damschroder, L. (2007). Qualitative Content Analysis (pp. 39-62). https://doi.org/10.1016/S1479-3709(07)11003-7
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Landsverk, J., Brown, C. H., Smith, J. D., Chamberlain, P., Curran, G. M., Palinkas, L., … McCue Horwitz, S. (2018). Design and Analysis in Dissemination and Implementation Research. In: Lewis, C. C., Proctor, E. K., & Brownson, R. C. (Eds.). Measurement Issues in Dissemination and Implementation Research (pp.201-227). Oxford University Press.
- [Background] Mayring, P. (2014). Qualitative Content Analysis Theoretical Foundation, Basic Procedures and Software Solution. Retrieved from http://nbn-resolving.de/urn:nbn:de:0168-ssoar-395173
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Squires, J. E., Hutchinson, A., Hayduk, L., Cranley, L. A., Cummings, G., Norton, P. G., & Estabrooks, C. A. (2014). Alberta Context Tool User Manual 2014.
- [Background] Stevens BJ, Yamada J, Estabrooks CA, Stinson J, Campbell F, Scott SD, Cummings G; CIHR Team in Children's Pain. Pain in hospitalized children: Effect of a multidimensional knowledge translation strategy on pain process and clinical outcomes. Pain. 2014 Jan;155(1):60-68. doi: 10.1016/j.pain.2013.09.007. Epub 2013 Sep 8. PMID 24021861
- [Background] Stevens BJ, Yamada J, Promislow S, Stinson J, Harrison D, Victor JC; Members of the CIHR Team in Children's Pain. Implementation of multidimensional knowledge translation strategies to improve procedural pain in hospitalized children. Implement Sci. 2014 Nov 25;9:120. doi: 10.1186/s13012-014-0120-1. PMID 25928349
- [Background] Tariman JD, Berry DL, Halpenny B, Wolpin S, Schepp K. Validation and testing of the Acceptability E-scale for web-based patient-reported outcomes in cancer care. Appl Nurs Res. 2011 Feb;24(1):53-8. doi: 10.1016/j.apnr.2009.04.003. Epub 2009 Sep 18. PMID 20974066
- [Derived] Stevens B, Bueno M, Barwick M, Campbell-Yeo M, Chambers C, Estabrooks C, Flynn R, Gibbins S, Harrison D, Isaranuwatchai W, LeMay S, Noel M, Stinson J, Synnes A, Victor C, Yamada J. The implementation of infant pain practice change resource to improve infant procedural pain practices: a hybrid type 1 effectiveness-implementation study. Pain. 2024 Dec 6;166(7):1587-1596. doi: 10.1097/j.pain.0000000000003496. PMID 39679622
- [Derived] Bueno M, Stevens B, Barwick MA, Riahi S, Li SA, Lanese A, Willan AR, Synnes A, Estabrooks CA, Chambers CT, Harrison D, Yamada J, Stinson J, Campbell-Yeo M, Noel M, Gibbins S, LeMay S, Isaranuwatchai W. A cluster randomized clinical trial to evaluate the effectiveness of the Implementation of Infant Pain Practice Change (ImPaC) Resource to improve pain practices in hospitalized infants: a study protocol. Trials. 2020 Jan 6;21(1):16. doi: 10.1186/s13063-019-3782-9. PMID 31907017